CLINICAL TRIAL: NCT04803188
Title: A Randomized Controlled Trial on the Role of Magnetic Resonance Imaging for Prostate Cancer Screening
Brief Title: Prostate Cancer Secondary Screening in Sapienza and Policlinico Umberto I
Acronym: ProSa-I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Valeria Panebianco, Professor of Radiology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5996
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: Prostate Cancer; Screening; Non-contrast MRI
MeSH Terms: conditions — Prostatic Neoplasms; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: patients will perform non-contrast MRI (Experimental): A: 355 patients will perform non-contrast MRI regardless their serum PSA value
  Interventions: Diagnostic Test: Magnetic Resonance
- B: patients will perform non-contrast MRI (Experimental): B: 355 patients will perform non-contrast MRI when serum PSA value is increased (>4 ng/ml or 2.5 ng/ml if positive family history)
  Interventions: Diagnostic Test: Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance — Screening MRI examinations will be performed on an MRI General Electric (GE) 3 Tesla MRI using a 32-channel phased array pelvic coil. The imaging protocol will include: T2-weighted morphological and diffusion-weighted functional sequences.
  All images will be reviewed by two radiologists experienced in urogenital imaging, who will be blinded to the patients' medical history. Both radiologists in charge will then assign a PI-RADS score (1 to 5) to each lesion for bi-parametric MRI, representing the likelihood of a clinically significant prostate lesion. For the generation of the overall PI-RADS score assigned to each lesion, the PI-RADS score algorithm for non-contrast MRI described in the PI-RADS version 2.1 recommendations will be applied. Lesions scored as bPI-RADS superior or equal than 3 will be directed to MRI-TRUS guided targeted biopsy.

SUMMARY:
Prostate Cancer (PCa) screening is still a controversial topic in the urology community, this is mostly linked to the low specificity of Prostate Specific Antigen (PSA) value. Screening with total PSA value has cause overdiagnosis of clinically insignificant prostate cancer (ciPCa) for many years, with lack of survival improvement. Non-contrast MRI, on the other hand, has become one of the most promising MRI applications, as it is a more sensitive test able to perform clinically significant PCa early detection. With this background the primary endpoint was to investigate the role of non-contrast MRI (without injection of paramagnetic contrast medium), as a secondary prevention test for the early diagnosis of prostate cancer, comparing it with the serum PSA test, in a randomized fashion.

DETAILED DESCRIPTION:
ENDPOINTS Primary endpoint To investigate the role of non-contrast Magnetic Resonance Imaging (MRI), as a secondary prevention test for the early diagnosis of prostate cancer (PCa), comparing it with the serum PSA test.

Secondary endpoints

1. Assess the percentage of men with a positive PSA screening test, defined as > 4 ng/ml and > 2.5 ng/ml in patients with family history of PCa (father and/or sibling).
2. Evaluation of the percentage of men with positive MRI and MRI targeted biopsy results stratified according to: absence of neoplasm, non-clinically significant neoplasm (ISUP 1) and clinically significant neoplasm (ISUP> 1), compared with PSA test and serum biomarkers (optional).
3. Comparison of the percentages of participants with PCa and with clinically significant PCa, according to the different positive screening tests.
4. Comparison of the different screening tests combinations in terms of PCa detection rate, both for non-clinically significant and clinically significant cancer.

STUDY DESIGN

Design:

Single center, prospective, interventional randomized controlled trial Duration: 2 years Evaluation of the effectiveness of the primary outcome: the evaluation of the effectiveness non-contrast MRI for the PCa detection will be based on MRI-guided biopsy targeted on the areas described and classified as biparametric Prostate Imaging-Reporting and Data System (bPI-RADS) ≥3 (scored according to the biparametric evaluation).

The reference standard for the diagnosis of prostate cancer will be the Magnetic Resonance Imaging - Transrectal Ultrasound (MRI-TRUS) guided targeted biopsy, which will be performed at a maximum of 4 weeks from MRI.

In order to evaluate the diagnostic accuracy of non-contrast MRI the diagnostic performance variables (sensitivity, specificity, accuracy, positive and negative predictive value, area under the curve and receiver operating characteristic curves) will be calculated.

For the statistical analysis of the effectiveness, only those participants who have undergone prostate biopsy as planned by the operator will be included.

In addition, the interreader agreement between two radiologists responsible for the analysis of MRI images, with 10 and 8 years of experience in urogenital imaging, respectively, will be evaluated. The agreement between the two radiologists will be calculated using the weighted Cohen's k statistic.

Evaluation of secondary outcomes: the evaluation of the effectiveness of secondary outcomes will be verified by evaluating the same statistical variables of diagnostic accuracy implemented for the primary purpose.

Safety evaluation: the safety of the procedure will be determined by assessing the incidence and severity of adverse events, defined as complications related to the procedure recorded from the first treatment and during the entire duration of the follow-up (2 years).

Participants in the study:

Enrollment: 710 men will be enrolled and blindly randomized in two different arms. Arm a) 355 patients will perform MRI with a bi-parametric approach (without contrast medium) regardless their PSA value; Arm b) 355 patients will perform MRI with a bi-parametric approach (without contrast medium) only when PSA is elevated.

Patients with positive MRI defined as bPI-RADS ≥3, will undergo MRI-directed targeted prostate biopsy.

ELIGIBILITY:
Inclusion criteria:

* Males aged between 49-69 years (from the age of 40 for those with family history of prostate cancer) at the time of enrollment
* Life expectancy greater than or equal to 10 years
* Sufficient understanding of the Italian language for written and verbal understanding of the information for enrollment in the Trial and for the process of obtaining informed consent.
* Patient with the ability to understand and want, able to express informed consent and to perform all the visits and procedures required by the study

Exclusion criteria:

* General contraindications to MRI
* Previous history of prostate cancer, prostate biopsy or treatment for prostate cancer
* Any contraindications to prostate biopsy, such as severe coagulation abnormalities (INR> 1.5), active urinary tract infection and acute prostatitis (NIH category I, II and III).
* Dementia or altered mental status that would prohibit understanding or granting informed consent

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 710 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of prostate cancer with non-contrast MRI | 24 months
  To investigate the role of MRI with a bi-parametric approach (without injection of paramagnetic contrast medium), as a secondary prevention test for the early diagnosis of prostate cancer, comparing it with the serum PSA test.

SECONDARY OUTCOMES:
Percentage of men with a positive PSA screening test | 2 years
  To assess the percentage of men with a positive PSA screening test, defined as > 4 ng/ml and > 2.5 ng/ml in patients with family history of prostate cancer (father and/or sibling).

OTHER OUTCOMES:
Stratification according to outcome | 2 years
  To evaluate the percentage of men with positive non-contrast MRI stratified according to: absence of neoplasm, non-clinically significant neoplasm (ISUP 1) and clinically significant neoplasm (ISUP> 1), compared with the tests of the PSA and serum biomarkers (optional).
Comparison of different positive screening tests | 2 years
  Comparison of the percentages of participants with the different positive screening tests. Comparison of the same in the subpopulation of patients with clinically significant neoplasia (ISUP> 1).
Comparison of different combination of screening tests | 2 years
  Comparison of the different combination of screening tests in terms of detection rate, non-clinically significant and clinically significant cancer detection rate.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Panebianco, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: Starting in January 2022, will be available for 6 months after publication
Access Criteria: The access will be granted to any researcher who will contact the principal investigator via email, upon reasonable request

REFERENCES:
- [Result] Epstein JI, Egevad L, Amin MB, Delahunt B, Srigley JR, Humphrey PA; Grading Committee. The 2014 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma: Definition of Grading Patterns and Proposal for a New Grading System. Am J Surg Pathol. 2016 Feb;40(2):244-52. doi: 10.1097/PAS.0000000000000530. PMID 26492179
- [Result] Matoso A, Epstein JI. Defining clinically significant prostate cancer on the basis of pathological findings. Histopathology. 2019 Jan;74(1):135-145. doi: 10.1111/his.13712. PMID 30565298
- [Result] Mottet N, van den Bergh RCN, Briers E, Van den Broeck T, Cumberbatch MG, De Santis M, Fanti S, Fossati N, Gandaglia G, Gillessen S, Grivas N, Grummet J, Henry AM, van der Kwast TH, Lam TB, Lardas M, Liew M, Mason MD, Moris L, Oprea-Lager DE, van der Poel HG, Rouviere O, Schoots IG, Tilki D, Wiegel T, Willemse PM, Cornford P. EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer-2020 Update. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2021 Feb;79(2):243-262. doi: 10.1016/j.eururo.2020.09.042. Epub 2020 Nov 7. PMID 33172724
- [Result] Welch HG, Albertsen PC. Reconsidering Prostate Cancer Mortality - The Future of PSA Screening. N Engl J Med. 2020 Apr 16;382(16):1557-1563. doi: 10.1056/NEJMms1914228. No abstract available. PMID 32294352
- [Result] Wegelin O, Exterkate L, van der Leest M, Kummer JA, Vreuls W, de Bruin PC, Bosch JLHR, Barentsz JO, Somford DM, van Melick HHE. The FUTURE Trial: A Multicenter Randomised Controlled Trial on Target Biopsy Techniques Based on Magnetic Resonance Imaging in the Diagnosis of Prostate Cancer in Patients with Prior Negative Biopsies. Eur Urol. 2019 Apr;75(4):582-590. doi: 10.1016/j.eururo.2018.11.040. Epub 2018 Dec 3. PMID 30522912
- [Result] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Result] Nam RK, Wallis CJ, Stojcic-Bendavid J, Milot L, Sherman C, Sugar L, Haider MA. A Pilot Study to Evaluate the Role of Magnetic Resonance Imaging for Prostate Cancer Screening in the General Population. J Urol. 2016 Aug;196(2):361-6. doi: 10.1016/j.juro.2016.01.114. Epub 2016 Feb 13. PMID 26880413
- [Result] Boesen L, Norgaard N, Logager V, Balslev I, Bisbjerg R, Thestrup KC, Winther MD, Jakobsen H, Thomsen HS. Assessment of the Diagnostic Accuracy of Biparametric Magnetic Resonance Imaging for Prostate Cancer in Biopsy-Naive Men: The Biparametric MRI for Detection of Prostate Cancer (BIDOC) Study. JAMA Netw Open. 2018 Jun 1;1(2):e180219. doi: 10.1001/jamanetworkopen.2018.0219. PMID 30646066
- [Result] Jambor I, Bostrom PJ, Taimen P, Syvanen K, Kahkonen E, Kallajoki M, Perez IM, Kauko T, Matomaki J, Ettala O, Merisaari H, Kiviniemi A, Dean PB, Aronen HJ. Novel biparametric MRI and targeted biopsy improves risk stratification in men with a clinical suspicion of prostate cancer (IMPROD Trial). J Magn Reson Imaging. 2017 Oct;46(4):1089-1095. doi: 10.1002/jmri.25641. Epub 2017 Feb 6. PMID 28165653
- [Result] Knaapila J, Jambor I, Ettala O, Taimen P, Verho J, Perez IM, Kiviniemi A, Pahikkala T, Merisaari H, Lamminen T, Saunavaara J, Aronen HJ, Syvanen KT, Bostrom PJ. Negative Predictive Value of Biparametric Prostate Magnetic Resonance Imaging in Excluding Significant Prostate Cancer: A Pooled Data Analysis Based on Clinical Data from Four Prospective, Registered Studies. Eur Urol Focus. 2021 May;7(3):522-531. doi: 10.1016/j.euf.2020.04.007. Epub 2020 May 14. PMID 32418878
- [Result] Eldred-Evans D, Burak P, Connor MJ, Day E, Evans M, Fiorentino F, Gammon M, Hosking-Jervis F, Klimowska-Nassar N, McGuire W, Padhani AR, Prevost AT, Price D, Sokhi H, Tam H, Winkler M, Ahmed HU. Population-Based Prostate Cancer Screening With Magnetic Resonance Imaging or Ultrasonography: The IP1-PROSTAGRAM Study. JAMA Oncol. 2021 Mar 1;7(3):395-402. doi: 10.1001/jamaoncol.2020.7456. PMID 33570542
- [Result] Panebianco V, Barchetti G, Simone G, Del Monte M, Ciardi A, Grompone MD, Campa R, Indino EL, Barchetti F, Sciarra A, Leonardo C, Gallucci M, Catalano C. Negative Multiparametric Magnetic Resonance Imaging for Prostate Cancer: What's Next? Eur Urol. 2018 Jul;74(1):48-54. doi: 10.1016/j.eururo.2018.03.007. Epub 2018 Mar 19. PMID 29566957
- [Result] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975